CLINICAL TRIAL: NCT02851628
Title: The Evaluation of an Alternative Sizing Model in Comparison of a Conventional Sizing Model for Full-face Masks in the Treatment of OSA in Terms of Performance and Comfort
Brief Title: The Evaluation of an Alternative Sizing Model in Comparison of a Conventional Sizing Model for Full Face Masks in the Treatment of OSA in Terms of Performance and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIA-194
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative sizing model trial mask (Experimental): In this arm participants who are randomized to the alternative sizing model based mask will be given the alternative sizing model based mask to use in home for the duration of this arm.
  Interventions: Device: Alternative sizing model based trial mask
- Prototype Full Face Mask (PFFM) (Active Comparator): In this arm, participants who are randomized to the PFFM will be given the PFFM to use in-home for the duration of this arm.
  Interventions: Device: Prototype Full Face Mask

INTERVENTIONS:
Device: Alternative sizing model based trial mask — A trial full face mask to be used for this trial for the treatment of obstructive sleep apnea using CPAP therapy.
  Arms: Alternative sizing model trial mask
Device: Prototype Full Face Mask — A prototype full face mask with previous clinical trial experience used for the treatment of obstructive sleep apnea using CPAP therapy.
  Arms: Prototype Full Face Mask (PFFM)

SUMMARY:
The investigation is a prospective non-blinded and semi-randomized clinical investigation. The investigation is designed to assess the alternative sizing model which the trial mask concept is based on and how it compares to a conventional sizing present in the Prototype Full Face Mask (PFFM) mask.

DETAILED DESCRIPTION:
The investigation is a prospective non-blinded and semi-randomized investigation. The investigation is designed to assess the alternative sizing model which the trial mask concept is based on and how it compares to a conventional sizing present in the Prototype Full Face Mask (PFFM) mask. A cohort of up to 38 pre-determined current nasal and full face mask users will be recruited by Fisher & Paykel Healthcare in Auckland New Zealand, Waikato DHB in Hamilton New Zealand, Hawkes Bay DHB in Hastings New Zealand and WellSleep Centre in Wellington New Zealand.

The study will involve baseline (visit one) gathering the participants' prescribed PAP therapy pressure and their usual mask (to have up-to-date records). The next visit (visit 2) 7 ± 4 days after visit 1, the participants will be fit the Prototype Full Face Mask (PFFM) mask or the alternative sizing based trial mask. At visit 3, which will be after 7 ± 4 days from visit 2, the participants will be crossed over to the mask. At visit 4, 7 ± 4 days after visit 3, all masks and devices will be collected from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give consent
* Apnea Hypopnea Index (AHI) ≥ 5 on diagnostic night
* Prescribed a Continuous Positive Airway Pressure (CPAP) device after successful OSA diagnosis
* Existing nasal or full face mask user.

Exclusion Criteria:

* Inability to give consent
* Patients who are in a coma or a decreased level of consciousness.
* Anatomical or physiological conditions making APAP therapy inappropriate (e.g. unconsolidated facial structure)
* Commercial drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of CO2 retention
* Pregnant or may think they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Seal Comfort | Up to 3 weeks in-home
  Obtained from subjective questionnaire
Subjective Seal Leak | Up to 3 weeks in-home
  Obtained from subjective questionnaire
Objective Seal Leak | Up to 3 weeks in-home
  Measured by device data

SECONDARY OUTCOMES:
Objective correct mask selection | Up to 3 weeks in-home
  Measured by device leak data
Subjective correct mask selection | Up to 3 weeks in-home
  Measured by subjective questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kayan Gonda, BSc, Principal Investigator — Sponsor Employee
Locations (4):
- New Zealand (4):
  - Hastings Memorial Hospital, Hastings, Hawkes Bay
  - Waikato Hospital (Waikato DHB), Hamilton, Waikato Region
  - Fisher & Paykel Healthcare, Auckland
  - Bowen Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No
This is a pilot investigation from which data will be used to inform product development on future projects and investigations.